CLINICAL TRIAL: NCT07239830
Title: Reference Values Determination of Nasal and Blood Interferon Scores in Uninfected Older Subjects REFérence Interféron Older Subjects (Older People Interferon Reference) - REFIPA Study
Brief Title: Interferon Reference for Older People - REFIPA Study
Acronym: REFIPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL25_0689
Record Dates: First submitted 2025-10-02; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Immunosenescence; Uninfected Older
Keywords: respiratory viral infection; Type I Interferon response; Older People; host-based response diagnostic test

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative and monocentric study, corresponding to researches involving human subjects (RIPH) category 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uninfected older adults (Other): Uninfected adult subjects aged 80 years and older
  Interventions: Other: Uninfected older adults

INTERVENTIONS:
Other: Uninfected older adults — The procedures specifically carried out for the study during a single visit are as follows:
  * 1 nasopharyngeal swab for baseline measurement of nasal IFN score and testing for infection
  * Venous blood sampling on:
    * 1 x 2 mL Paxgene tube for baseline measurement of blood IFN score
    * 3 x 10 mL EDTA tubes for collection of PBMCs and plasma to quantify anti-IFN antibody levels and lymphocyte subtype concentrations.
  A total of 32 mL of venous blood will be collected for the study during a single visit.
  A biological collection will be created with the participant's specific consent, using leftover blood and nasopharyngeal swabs after testing.

SUMMARY:
The diagnosis of respiratory viral infections is mainly based on PCR tests targeting the DNA or RNA of suspected viruses, including SARS-CoV-2, RSV and influenza viruses. However, this method is limited because it only tests for a small number of viruses, while many other pathogens can cause similar symptoms. As a result, respiratory viral infections are often underdiagnosed because not all possible viruses are systematically tested for.

Another limitation of PCR tests is that they can detect residual viral genetic material long after the infection has ended, making it difficult to distinguish between an active infection and a past one. Viral load can help interpret the result, but it is not always reliable. It is therefore essential to have complementary markers that can indicate whether the detected virus is still in the active replication phase.

An innovative approach is to measure the host's immune response, in particular the production of type I interferons (IFN-I), which are markers of active viral infection. Studies have shown that joint analysis of the IFN-I/III response and PCR tests improves the detection of viral respiratory infections by better discriminating between active infections. This method shows promise for refining diagnosis, particularly in cases where the viral load is low or ambiguous.

These advances are particularly important for older patients, in whom viral infections have a severe impact. Ageing leads to a decline in immune function (immunosenescence), including a reduction in IFN-I production. This alteration could further complicate the interpretation of immune biomarkers in older people, highlighting the need to establish reference values specific to this population.

In this context, the RESPIGERIA study (compliance with MR004 No. 24-5127) was launched to evaluate the IFN response in geriatric hospitalised patients with respiratory viral infections. However, there is still a lack of reference data on the IFN response in uninfected older individuals. Establishing a baseline IFN score in this population is essential in order to adapt diagnostic tools to age-related specificities.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 80 or over
* Patient admitted to the Charpennes hospital day unit or outpatient clinic for follow-up OR accompanying patient who receive care at the Charpennes geriatric hospital OR subject recruited through the local press
* Weight greater than or equal to 45 kg
* Subject living in the Lyon metropolitan area

Exclusion Criteria:

* Subjects with symptoms of active infection (symptom questionnaire or temperature > 37.5°C).
* Subjects with an autoimmune disease linked to a dysregulated interferon response.
* Subjects participating in another interventional study involving an exclusion period that is still ongoing or that may interfere with the present protocol.
* Subjects deprived of their liberty by judicial or administrative decision
* Subjects receiving psychiatric care
* Adults subject to legal protection measures (guardianship, curatorship)
* Subjects not affiliated with a social security scheme or beneficiaries of a similar scheme

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Nasal IFN-I scores measurement in a non-infected geriatric population. | The primary outcome will be measured at inclusion visit only
  IFN-I score will be measured by assessing the expression of a selection of IFN-I-stimulated genes.
Blodd IFN-I scores measurement in a non-infected geriatric population. | The primary outcome will be measured at inclusion visit only
  IFN-I score will be measured by assessing the expression of a selection of IFN-I-stimulated genes.

SECONDARY OUTCOMES:
Correlation between clinical parameters assessed by the Charlson score (comorbidities) and the Fried phenotype (frailty), and the basal blood and nasal interferon score | The secondary outcome will be measured at inclusion visit only
  We hypothesize that frailty (assessed by Frailty phenotype) and comorbidities (assessed by Charlson comorbidity index) could be associated with immunosenescence and IFN-I score.
Correlation between immune parameters assessed by anti-IFN antibody concentration, concentration of lymphocyte subtypes expressing or not expressing exhaustion markers (Tim-3, PD-1, etc.) and basal blood and nasal interferon score. | The secondary outcome will be measured at inclusion visit only
  Spearman correlation will be done between IFN-I score and each immune parameters.
Measurement of nasal IFN-I scores in a population of uninfected vs. infected older individuals (RESPIGERIA study, compliance with MR004 No. 24-5127). | The secondary outcome will be measured at inclusion visit only
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (uninfected vs. infected older individuals).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes (Hospices Civils de Lyon), Villeurbanne, France